CLINICAL TRIAL: NCT04267029
Title: Transfusion-Associated Dyspnea: Prospective Observational and Laboratory Assessment
Brief Title: Transfusion Associated Dyspnea Profiling
Acronym: TADPOL
Status: Completed | Type: Observational
Sponsor: Toronto Transfusion Medicine Collaborative (Other)
Collaborators: University Health Network, Toronto (Other); Sunnybrook Health Sciences Centre (Other); MOUNT SINAI HOSPITAL (Other); Unity Health Toronto (Other); Canadian Blood Services (Other)
Responsible Party: Sponsor
Other Study IDs: TADPOL_v0.7
Record Dates: First submitted 2020-02-07; First posted 2020-02-12 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Transfusion Reaction
Keywords: TACO (transfusion associated circulatory overload); TRALI (transfusion related acute lung injury); Allergic Reaction; FNHTR (febrile non-hemolytic transfusion reaction); TAD (transfusion associated dyspnea)
MeSH Terms: conditions — Transfusion Reaction; Transfusion-Related Acute Lung Injury; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Post-reaction plasma and serum and cellular pellets Implicated blood product residua
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: CRTR (cardiorespiratory transfusion reaction): Respiratory/cardiovascular disturbances after transfusion (>/=2 of respiratory distress, pulmonary edema, cardiovascular system changes, fluid shifts, cardiac strain indicators), with or without accompanying (or pre-existing) fever
  Interventions: Diagnostic Test: TADPOL battery (deep clinicolaboratory profile)
- Controls: HRFTR (high risk febrile transfusion reactions): Post-transfusion fevers requiring laboratory investigation (Tmax>/=39C, or lesser deflections if accompanied by chills/rigors), without respiratory features (hypoxia or dyspnea)
  Interventions: Diagnostic Test: TADPOL battery (deep clinicolaboratory profile)

INTERVENTIONS:
Diagnostic Test: TADPOL battery (deep clinicolaboratory profile) — profile dimensions:
  * hemolytic
  * allergic
  * cardiorenal
  * inflammatory
  * leukoagglutinating
  * exploratory bioarchive

SUMMARY:
Transfusion reactions are defined as harms occurring during or after blood transfusion, with new heart/lung stress (eg. troubled breathing) regarded as cardiorespiratory transfusion reactions (CRTRs). CRTRs are among the most important, as the leading cause of transfusion-related harm and death. Though there are distinct classifications for these events, real life cases often don't fall neatly into a given category, with outliers regarded as "transfusion associated dyspnea (TAD)". It is unknown what TAD is -- whether it has a unique root cause, is a milder version of other known CRTRs, or is a blend of events. The purpose of this study is to better understand TAD and CRTRs by profiling them through a detailed medical history and more intensive laboratory assessment. This review of CRTRs may improve the quality/validity of final conclusions reported in the health record and to hemovigilance bodies, and uncover the nature of TAD and/or minimize CRTRs defaulting to the TAD category. Our enhanced understanding will advance diagnostic, treatment, and prevention efforts.

DETAILED DESCRIPTION:
"Transfusion-Associated Dyspnea: Prospective Observation and Laboratory Assessment" (TADPOL) aims to improve the diagnosis and characterization of cardiorespiratory transfusion reaction (CRTR) patients ("cases"), as compared with high risk febrile transfusion reaction (HRFTR) patients ("controls"), by applying a standardized and intensive clinicolaboratory profiling tool.

CRTR, in contrast with HRFTR, are more difficult to diagnose and manage. Patients are often sick with (or prone to) pathologies that resemble reactions (eg. congestive heart failure [CHF] vs transfusion associated circulatory overload [TACO]), and/or experience more than one transfusion-associated disturbance at a time.

CRTRs are also the most disruptive, distressing, and disposition-escalating events for patients at an individual level, and are disproportionately accountable for transfusion associated deaths at the collective level in national hemovigilance systems. The cardinal CRTRs range from TACO (most commonly) to allergic bronchospasm to transfusion related acute lung injury (TRALI).

Inaccurate classification may undercount certain phenomena (when criteria fail to be met by confounding conditions), and/or overcount others (when including all possibilities-of-relevance in hemovigilance).

These uncertainties beget gaps (or excesses) in patient care and in donor/product-associated decision-making.

HYPOTHESES: The TADPOL CRF and laboratory profiling effort will improve the yields of confident (more certain), accurate (better-grounded), and thorough (multi-event-sensitive) diagnoses in CRTR patients.

Most cases of TAD are likely to be re-classified as milder versions (or overlaps) of possible CRTR states (± the underlying condition), while the remainder may exhibit a signature resembling FNHTR (FTR controls).

Precise case-mapping should yield useful personalized information, while aggregated findings from each disturbance pathway - as they are distributed in each conventional reaction category - can validate the utility of markers being explored in reaction investigation algorithms.

The TADPOL bioarchive and anonymized dataset will also be assets for explorations of novel indicators and patterns.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Transfusion of blood products (components or derivatives) with an available pre-transfusion group & screen specimen
* Referred to the blood transfusion laboratory for review of a suspected acute transfusion reaction (occurring within 24 hours of completing transfusion), and either exhibiting a cardiorespiratory disturbance (CRTR: cases) or a high-risk febrile disturbance (HRFTR: controls)

Exclusion Criteria:

* Pregnant females
* Massive hemorrhage entailing >20 implicated products in the 24h period before the acute transfusion reaction's onset
* Previous enrolment in the same designation (ie- an individual with RTR will not re-enroll if having another RTR, but may re-enrol if having FTR)
* Expected to discharge home or die sooner than specimen acquisition
* Withdrawal of consent at any time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients at 4 university-affiliated teaching hospitals who have received a blood transfusion, and experienced a suspected acute transfusion reaction
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
CERTAINTY | 2 years
  Improve certainty in final cardiorespiratory transfusion reaction event classifications (by reduction in the number of cases otherwise achieving no better than "possible" provisional conclusions), from the expected base ambiguity rate of 60%, down to 30%.

SECONDARY OUTCOMES:
COMPLEXITY | 2 years
  Determine the frequency of multi-domain disturbances (ie- "overlap") in cardiorespiratory transfusion reaction referrals
PATHOGENESIS FOOTPRINTING | 2 years
  Statistically characterize concordance of established and potential criteria in TRALI, TACO, allergic bronchospasm, and TAD

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Csert-Gazdewich, MD, Principal Investigator — Universith Health Network
Locations (4):
- Canada (4):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Callum JL, Cohen R, Cressman AM, Strauss R, Armali C, Lin Y, Pendergrast J, Lieberman L, Scales DC, Skeate R, Ross H, Cserti-Gazdewich C. Cardiac stress biomarkers after red blood cell transfusion in patients at risk for transfusion-associated circulatory overload: a prospective observational study. Transfusion. 2018 Sep;58(9):2139-2148. doi: 10.1111/trf.14820. PMID 30204946
- [Background] Cohen R, Escorcia A, Tasmin F, Lima A, Lin Y, Lieberman L, Pendergrast J, Callum J, Cserti-Gazdewich C. Feeling the burn: the significant burden of febrile nonhemolytic transfusion reactions. Transfusion. 2017 Jul;57(7):1674-1683. doi: 10.1111/trf.14099. Epub 2017 Mar 28. PMID 28369916
- [Background] Parmar N, Pendergrast J, Lieberman L, Lin Y, Callum J, Cserti-Gazdewich C. The association of fever with transfusion-associated circulatory overload. Vox Sang. 2017 Jan;112(1):70-78. doi: 10.1111/vox.12473. Epub 2016 Dec 21. PMID 28001310
- [Background] McVey MJ, Cohen R, Arsenault V, Escorcia A, Tasmin F, Pendergrast J, Lieberman L, Lin Y, Callum J, Cserti-Gazdewich C. Frequency and timing of all-cause deaths in visits involving suspected transfusion reactions, and the significance of cardiopulmonary disturbances. Vox Sang. 2021 Sep;116(8):898-909. doi: 10.1111/vox.13086. Epub 2021 Feb 26. PMID 33634884
- See also: TADPOL Protocol paper — https://ijclinicaltrials.com/index.php/ijct/article/view/645